CLINICAL TRIAL: NCT04778241
Title: Effects of Mini Implant Facilitated Micro-osteoperforations on the Alignment of Mandibular Anterior Crowding: A Randomized Controlled Clinical Trial
Brief Title: Effects of Mini Implant Facilitated Micro-osteoperforations on the Alignment of Mandibular Anterior Crowding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Assistant professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOP76
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Tooth Position Anomalies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding to treatment allocation was possible only for the investigator and data analyst because the clinicians could know the intervention as osteo-perforation can be obviously seen clearly. Masking the intervention for the participants were not possible because micro-osteoperforation is a surgical procedure. All the trial documents were labeled with the study ID number, which was used for participant identification and data collection without unmasking the allocation group. This allowed the investigator to complete data collection and measurements blindly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-Osteoperforation group (Experimental): All the participants bonded by the care provider with 0.022 inch MBT prescription appliance (Ortho TechanologyTM,USA). Mini-implant facilitated micro-osteoperforation (MOPs) were placed in the experimental group before placing the initial leveling arch wire. MOPs were placed at three sites i.e., interproximally between mandibular canine and lateral incisor on both sides and between central incisors in the midline on labial aspect of mandible.
  Interventions: Procedure: Micro-osteoperforation
- Control group (No Intervention): All the participants in this group bonded by the principal investigator with 0.022-inch slot MBT prescription appliance (Ortho TechanologyTM,USA). No micro-osteoperforation was used in this group.

INTERVENTIONS:
Procedure: Micro-osteoperforation — Mini-implant facilitated micro-osteoperforation (MOPs) were placed in the experimental group before placing the initial leveling arch wire. MOPs were placed at three sites i.e., interproximally between mandibular canine and lateral incisor on both sides and between central incisors in the midline on labial aspect of mandible.
  Other Names: MOP
  Arms: Micro-Osteoperforation group

SUMMARY:
The primary aim of the present study is to evaluate the the efficacy of micro-osteoperforation (MOPs) perfomed by mini-implant (MI) screw In improving alignment of mandibular anterior teeth

DETAILED DESCRIPTION:
Primarily the present study is designed to evaluate the efficacy of micro-osteoperation (MOPs) perfomed by mini-implant (MI) screw In improving alignment of mandibular anterior teeth. Additionally, the possibility of inducing root resorption, and patient perception of pain during the initial phase of treatment.

Subjects and Methods: Orthodontic patients aged 17-25 years old, non-extraction treatment with lower anterior crowding of 4-6 mm using Little's irregularity index. Outcome measures included the amount of crowding using Little's irregularity index (LII), apical root resorption, and pain perception. The effectiveness of alignment will be tested using t-test, while root resorption and pain perception will be tested by the Mann-Whitney U test, and Wilcoxon signed-rank test (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 17-25years
2. Non-extraction treatment in the mandibular arch
3. Presence of full complement of dentition from first molar to first molar
4. Mandibular anterior irregularity index between 4-6 mm
5. Patient with healthy periodontium and no attachment loss of >2 mm

Exclusion Criteria:

1. Previous orthodontic treatment
2. Presence of primary or missing permanent teeth in the mandibular anterior area
3. Medical problems that affect tooth movement.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Alignment efficiency | 4 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3D program (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.
Alignment efficiency | 8 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3D program (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.
Alignment efficiency | 12 weeks
  3D scanned study models were used to measure the amount of crowding in the mandibular anterior teeth using 3D program (DentalCad,Galway,3.0,2021). If Little's irregularity index is less than 1mm and alignment improvement not above 0.5 mm between two successive visits, then treatment is regarded as finished.

SECONDARY OUTCOMES:
The amount of Root resorption | 12 weeks
  The amount of root resorption was measured at the start of treatment and after 12 weeks, the length of the root was recoded at these time intervals. Radiographic films were positioned using a customized sensor holder for the lower anterior teeth with a 7cm film-cone distance using long cone paralleling technique. The radiographs were made at 70kV and 8mA DC with an exposure of 0.25 seconds.
Pain perception | first 7 days
  Evaluations of pain/discomfort was made in the evening on a daily basis over the first 7 days after bonding using a 10-point visual analog scale (VAS) of 10cm length. The highest pain level experienced should be reported by each patient. The recording sheet was received by all the patients on the day of bonding, it included seven visual analog scales (one for each day) and the patients were given oral instructions on how to finish the VAS by marking the point on the line which supposed to represent the maximum pain that they felt per day, with 0 refers to "no pain" and 10 refers to "intolerable pain". Patients were reminded daily by a phone call or a text message to mark the recording sheet and to bring it on their next appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Mushriq Abid, MSc, PhD, Principal Investigator — University of Baghdad
Locations (1):
- College of Dentisry-University of Baghdad, Baghdad, Iraq

REFERENCES:
- [Derived] Al-Attar A, Nissan L, Almuzian M, Abid M. Effect of mini-implant facilitated micro-osteoperforations on the alignment of mandibular anterior crowding: A randomised controlled clinical trial. J Orthod. 2022 Dec;49(4):379-387. doi: 10.1177/14653125221099038. Epub 2022 May 15. PMID 35575069